CLINICAL TRIAL: NCT06485180
Title: Women's Hospital, Zhejiang University School of Medicine
Brief Title: Comparative Effectiveness of Uterine Repair Surgery on Preventing Recurrence of Cesarean Sar Pregnancy
Acronym: CECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR02024-069
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: This retrospective study screened 1027 CSP individuals from the multiple center Medical Record Data System (MRDS) from three large hospitals in China, recorded between Jan 1, 2019, and Dec 31, 2022. 606 patients underwent surgical treatment. The pregnancy outcomes and contraceptive methods were all reviewed through telephone follow-up. Conservative surgeries included dilatation and curettage (D&C) and hysteroscopy and resection surgeries included CSP excision plus hysterotomy closure.
Who Masked: Outcomes Assessor
Masking Description: The pregnancy outcomes and contraceptive methods were all reviewed through telephone follow-up. All outcomes Assessor were provided patients' name and telephone without surgery methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative surgery (Active Comparator): D&C: A curette is inserted into the uterus through the dilated cervix. The curette is used to scrape the lining of the uterus and remove the pregnancy tissue.
  Hysteroscopy: The procedure can be used for CSP with progression toward the uterine cavity or the bladder. The gestational sac is dissected free of the uterine wall through a natural entrance, and hemostasis can be achieved with electro-coagulation using a wire-loop or roller-ball. Hysteroscopy is a minimally invasive technique and is conducted under direct observation or combined with abdominal ultrasound.
  Interventions: Procedure: Active comparator
- Resection surgery (Active Comparator): Transvaginal CSP excision: The bladder is dissected away through an incision in the anterior cervico-vaginal junction, and the CSP is identified in the anterior part of the lower uterine segment. The ectopic pregnancy tissue is removed through a transverse incision, and suction curettage through the incision on the uterus can be performed. Finally, the myometrial and vaginal defects are repaired.
  Hysteroscopy-assisted laparoscopic CSP excision: Under the guidance of the light of hysteroscopy, position CSP accurately and excision is performed of the uterine scar that contains the ectopic pregnancy, with subsequent repair of the defect in the uterus. After laparoscopic CSP excision, hysteroscopy proved that the niche had disappeared.
  Abdominal CSP excision: The ectopic pregnancy tissue is removed through an abdominal incision, and suction curettage through the incision on the uterus can be performed. Finally, the myometrial and abdominal defects are repaired.
  Interventions: Procedure: Active comparator

INTERVENTIONS:
Procedure: Active comparator — Participants from conservative group were selected as uterine curettage (D&C) cohort , hysteroscopy cohort, Uterine Artery Embolization (UAE) in Combination with D&C, without MTX cohort, UAE in Combination D&C with MTX cohort and UAE+ D&C+hysteroscopy.
  Participants from CSP excision plus hysterotomy closure group were selected as transvaginal CSP excision cohort, hysteroscopy-assisted laparoscopic CSP excision cohort and abdominal CSP excision cohort.

SUMMARY:
The goal of this observational study is to learn about the long-term effects of resection surgery which is cesarean scar pregnancy(CSP) excision plus hysterotomy closure in CSP patients to treat their CSP. The main question it aims to answer is:

Does resection surgery lower next recurrence of CSP than conservative surgery which leaves the uterine niche alone? Participants already underwent resection surgery or conservative surgery will answer survey questions about their next pregnancy for 3 years.

DETAILED DESCRIPTION:
Background Cesarean scar pregnancy (CSP) is a rare but prognostically severe obstetrics and gynecology complication. There have been well-developed techniques for the initial treatment of CSP. However, the recurrence of CSP remains a challenge for clinicians. Currently, the conservative surgery and resection surgery has been widely applied in clinical practice, However, there is no published data exist regarding whether hysterotomy closure technique for CSP can prevent recurrence of CSP. The investigators aimed to systematically evaluate the value of hysterotomy closure on the prevent on recurrent CSP and improve pregnancy outcome.

Methods In this multi-centre, retrospective cohort study, participants hospitalized three hospitals in China due to CSP from January 1, 2019 to December 31, 2022 were collected, and their pregnancy outcomes were followed up until January 31, 2024. International and Chinese classifications were determined based on the results of three-dimensional ultrasound. A total of 606 CSP patients who met the criteria were included in our analysis. Based on Chinese classification, 171 CSP I, 404 CSP II and 31 CSP III were identified. Based on international classification, 575 endogenous CSP and 31 exogenous CSP were identified. The investigators compared the baseline data of two groups of subjects regarding fertility, excluding cases with no fertility requirements or incomplete information. Effectiveness was used to compare the resection surgery and conservative surgery in clinical practice. Survival analysis was used to examine the relationship among post-surgical pregnancy interval and recurrent CSP. The primary outcome was the effectiveness which included successful termination of the current CSP and non-CSP in the next pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. This retrospective study screened 1027 CSP individuals from the multiple center Medical Record Data System (MRDS) from three large hospitals in China, recorded between Jan 1, 2019, and Dec 31, 2022.
2. Conservative surgeries included dilatation and curettage (D&C) and hysteroscopy, and resection surgeries included CSP excision plus hysterotomy closure
3. Based on the widespread clinical utility of diagnostic criteria, four factors pertaining to patients, namely amenorrhea, clinical manifestations, laboratory results, and 3-D ultrasound or MRI findings, were thoroughly examined.
4. All participants were subsequently verified pathologically to confirm the presence of CSP.
5. Chinese CSP classification was selected as investigate group.
6. The international group encompasses endogenous and exogenous were selected as control group.

Exclusion Criteria:

1. those with incomplete medical record information or follow-up data;
2. those who did not undergo their first surgery at any of the three hospitals;
3. individuals without fertility requirements or have adopted long-term contraception were excluded;
4. who underwent surgery after December 31, 2022 were excluded, even if they became pregnant during the follow-up time.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cesarean scar pregnancy can happened to female only.
Enrollment: 606 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
effectiveness | up to 3 years
  The incidence rate of non-CSP

CONTACTS AND LOCATIONS:
Overall Officials: Xiuxiu Jiang, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's hospital, school of medicine, zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No